CLINICAL TRIAL: NCT01737762
Title: A Phase 3 Randomized, Double Blind, Vehicle Controlled Study Investigating the Safety and Efficacy of HP802-247 in the Treatment of Venous Leg Ulcers >12 cm2 to ≤ 36 cm2
Brief Title: Study Investigating the Safety and Efficacy of HP802-247 in the Treatment of Venous Leg Ulcers >12 cm2 to ≤ 36 cm2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Healthpoint (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 802-247-09-031
Record Dates: First submitted 2012-11-20; First posted 2012-11-30 (Estimated); Results first posted 2017-07-26 (Actual); Last update posted 2017-07-26 (Actual); Status verified 2016-09

CONDITIONS: Venous Leg Ulcers
Keywords: Venous leg ulcer; ulcer; Venous stasis; compression; venous; venous stasis ulcer; vlu; wound; varicose veins; venous insufficiency; dvt; deep vein thrombosis
MeSH Terms: conditions — Varicose Ulcer; Ulcer; Wounds and Injuries; Varicose Veins; Venous Insufficiency; Venous Thrombosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HP802-247 (Experimental): HP802-247 (fibrinogen solution & thrombin solution containing living, irradiated, growth arrested keratinocytes and fibroblasts) 260 solution) containing 0.5 x 106 cells per mL every 14 days.
  Interventions: Biological: HP802-247
- Vehicle (Placebo Comparator): Vehicle Control(fibrinogen solution & thrombin solution without cells)
  Interventions: Biological: Vehicle

INTERVENTIONS:
Biological: HP802-247 — HP802-247 (fibrinogen solution & thrombin solution containing living, irradiated, growth arrested keratinocytes and fibroblasts) 260 µL (130 µL, one spray, of each solution) containing 0.5 x106 cells per mL every 14 days.
  Arms: HP802-247
Biological: Vehicle
  Arms: Vehicle

SUMMARY:
This study is being done to find out if an investigational product called HP802-247 can help people with venous leg ulcers. Investigational means that HP802-247 has not been approved by the U.S. Food and Drug Administration (FDA).

At least 250 subjects will participate. The study is going to be conducted in approximately 50 sites in the United States and Canada.

DETAILED DESCRIPTION:
This research is being done to compare the efficacy of HP802-247 plus compression therapy against Vehicle plus compression therapy in achieving complete wound closure over the 16-week treatment period. Vehicle looks the same as HP802-247 but contains no cells. Target wound status is evaluated at each study visit (closed, open, reopened). At wound closure or completion of treatment all subject will enter an observational safety followed up period which ends at one year after initial exposure to test article.

ELIGIBILITY:
Inclusion Criteria:

* Provide informed consent.
* Age ≥ 18 years and of either sex.
* Willing to comply with protocol instructions, including allowing all study assessments.
* Have a venous leg ulcer (VLU) between the knee and ankle (at or above the malleolus), with a surface area >12 cm2 to ≤ 36 cm2
* Venous insufficiency confirmed by duplex Doppler ultrasound examination for valvular or venous incompetence.
* Arterial supply adequacy confirmed
* Target ulcer involves a full thickness skin loss, but WITHOUT exposure of tendon, muscle, or bone.
* Target ulcer duration ≥ 6 weeks but ≤ 104 weeks (24 months).
* Acceptable state of health and nutrition

Exclusion Criteria:

* History of anaphylaxis, serum sickness, or erythema multiforme reaction to aprotinin, bovine serum albumin or bovine serum proteins, penicillin, streptomycin, amphotericin B.
* Prior diagnosis of Systemic Lupus Erythematosus with elevated anti-DNA antibody titers, Buerger's disease (thromboangiitis obliterans), current diagnosis of vasculitis, or current diagnosis of claudication.
* Therapy with another investigational agent within thirty (30) days of Screening, or during the study.
* A target ulcer of non-venous etiologies (e.g., sickle cell anemia, necrobiosis lipoidica diabeticorum, pyoderma gangrenosum, vasculopathic or vasculitic).
* Documented history of osteomyelitis at the target wound location within 6 months preceding the Screening Visit.
* Refusal of or inability to tolerate compression therapy.
* Therapy of the target ulcer with autologous skin graft, Apligraf™, or Dermagraft™ within 30 days preceding the Screening Visit.
* History of cancer in the preceding 5 years (other than carcinoma in situ of the cervix or adequately treated non-melanoma skin cancers).
* Any prior exposure to HP802-247 or its vehicle.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2012-11; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Herbert B Slade, MD, Study Chair — Healthpoint; Tommy Lee, MSHS, Study Director — Healthpoint; Robert Kirsner, MD, Principal Investigator — University of Miami; William Marston, MD, Principal Investigator — University of North Carolina
Locations (41):
- United States (35):
  - Phoenix, Arizona
  - Carlsbad, California
  - Castro Valley, California
  - Fair Oaks, California
  - Fresno, California
  - Laguna Hills, California
  - Long Beach, California
  - Los Angeles, California
  - San Diego, California
  - Sylmar, California
  - Washington D.C., District of Columbia
  - Hialeah, Florida
  - Miami, Florida
  - South Miami, Florida
  - Chicago, Illinois
  - Jacksonville, Illinois
  - Springfield, Illinois
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Saginaw, Michigan
  - Washington, Missouri
  - Las Vegas, Nevada
  - Bayonne, New Jersey
  - Hoboken, New Jersey
  - East Meadow, New York
  - New York, New York
  - Chapel Hill, North Carolina
  - Akron, Ohio
  - Willoughby, Ohio
  - Tulsa, Oklahoma
  - Dunmore, Pennsylvania
  - Wyomissing, Pennsylvania
  - Knoxville, Tennessee
  - Fort Worth, Texas
  - Tacoma, Washington
- Canada (5):
  - Calgary, Alberta
  - Winnipeg, Manitoba
  - Hamilton, Ontario
  - London, Ontario
  - Sherbrooke, Quebec
- San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
Results summaries have been sent to each site for distribution to participants

REFERENCES:
- [Derived] Marston WA, Ennis WJ, Lantis JC 2nd, Kirsner RS, Galiano RD, Vanscheidt W, Eming SA, Malka M, Cargill DI, Dickerson JE Jr, Slade HB; HP802-247 Study Group. Baseline factors affecting closure of venous leg ulcers. J Vasc Surg Venous Lymphat Disord. 2017 Nov;5(6):829-835.e1. doi: 10.1016/j.jvsv.2017.06.017. PMID 29037354

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were screened at 36 sites in the US and 3 in Canada; between November 30, 2012 and November 11, 2015; sites included independent and hospital wound clinics and private practice sites.
Pre-assignment Details: Subjects entered a 2-week run-in; subjects whose wound radius decreased by < 0.349 cm/2weeks and met all other inclusion/exclusion (I/E) criteria were eligible for randomization. After completion of the treatment period, subjects entered a three-month follow up period.
Period: Overall Study
Arm/Group | HP802-247 | Vehicle
Started | 77 | 78
Completed | 57 | 61
Not Completed | 20 | 17
Not completed — Adverse Event | 2 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Progressive disease | 1 | 2
Not completed — Physician Decision | 1 | 1
Not completed — Moved from area | 2 | 1
Not completed — Trial termination | 11 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HP802-247 | Vehicle | Total
Number analyzed (Participants) | 69 | 70 | 139
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 37 | 44 | 81
  >=65 years | 32 | 26 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.4 (15.1) | 61.0 (12.1) | 61.7 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 32 | 60
  Male | 41 | 38 | 79
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 15 | 32
  Not Hispanic or Latino | 52 | 55 | 107
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 11 | 24
  White | 51 | 58 | 109
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  Canada | 4 | 3 | 7
  United States | 65 | 67 | 132

OUTCOME MEASURES:

1. Primary Outcome: Wound Closure
Description: Compare HP802-247 plus compression therapy against Vehicle plus compression therapy for proportion of subjects with complete wound closure over the 16-week treatment period from baseline.
Time Frame: 16 Weeks
Measure: Number; unit: participants
Arm/Group | HP802-247 | Vehicle
Number analyzed (Participants) | 69 | 70
participants | 17 | 23

2. Secondary Outcome: Time in Days to Closure
Description: Compare the efficacy of HP802-247 plus compression therapy against Vehicle plus compression therapy in achieving complete wound closure, based on time in days to closure over the 16-week treatment period from baseline.
Time Frame: 16 Weeks
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | HP802-247 | Vehicle
Number analyzed (Participants) | 69 | 70
Days | 83.4 (33.8) | 87.1 (42.5)

ADVERSE EVENTS:
Time Frame: Treatment emergent Adverse Events (AE) were collected weekly during the 16-week treatment period; post treatment AE were collected during the follow up period.
Description: Adverse events were reported at each study visit over the duration of the study
Groups:
- Vehicle: Vehicle Control(fibrinogen solution & thrombin solution without cells)
  Vehicle
Arm/Group | HP802-247 | Vehicle
All-Cause Mortality (participants affected / at risk) | 0/77 | 0/78
Serious Adverse Events (participants affected / at risk) | 7/77 | 7/78
Other Adverse Events (participants affected / at risk) | 23/77 | 19/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HP802-247 (N=77) | Vehicle (N=78)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 2 (2) | 1 (1)
Infected skin ulcer (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Pulmonary embo;ism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Peripheral ischemia (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HP802-247 (N=77) | Vehicle (N=78)
Cellulitis (Infections and infestations) | 8 (9) | 5 (6)
Infected skin ulcer (Infections and infestations) | 2 (2) | 3 (3)
Wound infecton (Infections and infestations) | 3 (5) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 4 (5) | 4 (4)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 11 (17) | 8 (13)

LIMITATIONS AND CAVEATS:
The trial was terminated due to the failure of the Phase 3 study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less